CLINICAL TRIAL: NCT00988637
Title: An Open-label, Multi-center, Randomized, Evaluator-Blinded Study to Evaluate the Safety and Efficacy of Two Treatment Regimens Involving Vectical™ (Calcitriol) Ointment 3 µg/g and Clobex® (Clobetasol Propionate) Spray, 0.05% in the Treatment of Moderate Plaque Psoriasis
Brief Title: Evaluate Safety/Efficacy of Two Treatment Regimens for Vectical™ Ointment & Clobex® Spray for Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10144
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2012-09

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) Vectical™ Ointment and Clobex® Spray (Other): Vectical™ Ointment weekdays & Clobex® Spray weekends regimen
  Interventions: Drug: Vectical™ Ointment weekdays and Clobex® Spray weekends regimen
- 2) Clobex® Spray and Vectical™ Ointment (Other): Clobex® Spray morning and Vectical™ Ointment evening regimen
  Interventions: Drug: Clobex® Spray morning and Vectical™ Ointment evening regimen

INTERVENTIONS:
Drug: Vectical™ Ointment weekdays and Clobex® Spray weekends regimen — Vectical™ Ointment 3 µg/g, topical, apply twice daily on weekdays (Mon-Fri) and Clobex® Spray 0.05% twice daily on weekends (Sat-Sun) for 28 days
  Other Names: calcitriol ointment 3µg/g and clobetasol propionate spray 0.05%
  Arms: 1) Vectical™ Ointment and Clobex® Spray
Drug: Clobex® Spray morning and Vectical™ Ointment evening regimen — Clobex® Spray 0.05%, topical, apply once each morning and Vectical™ Ointment 3 µg/g, topical, apply once each evening for 28 days
  Other Names: clobetasol propionate spray 0.05% and calcitriol ointment 3 µg/g
  Arms: 2) Clobex® Spray and Vectical™ Ointment

SUMMARY:
This clinical trial will evaluate the efficacy and safety of Clobex® (clobetasol propionate) Spray 0.05% and Vectical™ (calcitriol) Ointment 3 µg/g over a four week period of use in one of two different regimens:

1. Vectical™ Ointment treatment, twice daily on weekdays (Mon - Fri) and Clobex® Spray treatment twice daily on weekends (Sat - Sun) for 28 days
2. Clobex® Spray once each morning and Vectical™ Ointment once each evening for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 80 years inclusive
* Subjects with an Overall Disease Severity of 3 (moderate)
* Subjects with 3% - 10% treatable BSA (Body Surface Area) excluding scalp, face, groin, axillae and/or other intertriginous areas
* For concurrent medications, type and dose must have been stable for at least 3 months prior to study entry and not expected to change during the study. Subjects receiving treatment with beta-blockers or lithium, whose dose has been stable for at lest 6 months and who have shown no worsening of their psoriasis, may be included in the study, at the discretion of the investigator

Exclusion Criteria:

* Subjects with intakes of more than 2,000 IU/day (50 mcg/day) of vitamin D (tolerable upper intake level) and/or more than 1,000 mg/day of calcium
* Subjects whose psoriasis involves only the scalp, face, groin, axillae, and/or other intertriginous areas
* Subjects with a wash-out period for topical treatment less than 30 days (Any steroid containing medication, dovonex, anthralin, tar and/or UVB treatment)
* Subjects with a wash-out period for systemic treatment less than 12 weeks (corticosteroids, biologics and/or PUVA treatment; Examples of these therapies include, but are not limited to PUVA, Soriatane, Cyclosporine, Hydroxyurea, Mycophenolate mofetil, Sulfasalazine, Azathioprine, Alefacept, Efalizumab, Adalimumab, Etanercept, Infliximab, Rituximab, and Methotrexate)
* Subjects with non-plaque psoriasis or other related diseases not classified as plaque psoriasis
* Subjects who foresee intensive UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (6):
- United States (5):
  - Dermatology Research Associates, Los Angeles, California
  - Therapeutics Clinical Research, San Diego, California
  - Hudson Dermatology, Evansville, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Baylor Research Institute Dermatology Research, Dallas, Texas
- Probity Medical Research, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Hudson CP, Kempers S, Menter A, Papp K, Smith S, Sofen H, Colon LE, Johnson LA, Gottschalk R. An open-label, multicenter study of the efficacy and safety of a weekday/weekend treatment regimen with calcitriol ointment 3 microg/g and clobetasol propionate spray 0.05% in the management of plaque psoriasis. Cutis. 2011 Oct;88(4):201-7. PMID 22106730
- [Derived] Menter A, Sofen H, Smith S, Papp K, Kempers S, Hudson CP, Colon LE, Johnson LA, Gottschalk R. An open-label, multicenter study of the efficacy and safety of an AM/PM treatment regimen with clobetasol propionate spray 0.05% and calcitriol ointment 3 microg/g in the management of plaque psoriasis. Cutis. 2011 Jul;88(1):46-51. PMID 21877508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on October 26, 2009 and the last subject was enrolled on January 28, 2010.
Pre-assignment Details: Wash-out period up to baseline is 30 days for any steroid containing medication, dovonex, anthralin, tar and/or ultraviolet B (UVB) treatment; 12 weeks for corticosteroids, biologics and/or psoralen + ultraviolet A (PUVA) treatment.
Groups:
- Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends): Vectical® Ointment, topical, apply twice daily on weekdays and Clobex® Spray, topical, apply twice daily on weekends for up to 28 days: Weekdays / Weekends Regimen
- Clobex® Spray (Morning) and Vectical® Ointment (Evening): Clobex® Spray, topical, apply once each morning and Vectical® Ointment, topical, apply once each evening for up to 28 days(PM): AM / PM Regimen
Period: Overall Study
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Started | 70 | 68
Completed | 67 | 65
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — non-compliance with study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening) | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (14.03) | 44.5 (14.43) | 45.4 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were a Success (Clear/Almost Clear) of Plaque Psoriasis at Week 4 Based on the Overall Disease Severity (ODS), Full Ordinal Scale From Baseline to Week 4
Description: Number of participants who were a success (Clear/Almost Clear) of Plaque Psoriasis at week 4 based on the Overall Disease Severity (ODS), full ordinal scale from baseline to week 4. Overall Disease Severity is evaluated on a scale from 0 - 4 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe/Very Severe) with 0 being best and 4 being worst.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants | 14 | 28

2. Secondary Outcome: Number of Participants Who Were a Success (Clear/Almost Clear) of Plaque Psoriasis at Week 2 Based on the Overall Disease Severity (ODS), Dichotomized Scale From Baseline to Week 2
Description: Number of participants who were a success (Clear/Almost Clear) of Plaque Psoriasis at Week 2 based on the Overall Disease Severity (ODS), dichotomized scale from Baseline to Week 2. Overall Disease Severity is evaluated on a scale from 0 - 4 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe/Very Severe) with 0 being best and 4 being worst.
Time Frame: Baseline to week 2
Population: ITT (Intent to Treat), LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants | 9 | 14

3. Secondary Outcome: Number of Participants in Each Category of the Global Assessment of Improvement (GAI) Scale From Baseline to Week 4
Description: Number of participants in each category of the Global Assessment of Improvement (GAI) Scale from Baseline to Week 4. The Global Assessment of Improvement is evaluated on a scale from -1 to 4 (-1 = Symptoms worse, 0 = No change, 1 = Minimal Improvement, 2 = Definite Improvement, 3 = Considerable Improvement and 4 = Clearing) with -1 being worst and 4 being best.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat); LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Symptoms worse (-1) | 1 | 0
  No change (0) | 2 | 6
  Minimal Improvement (1) | 9 | 6
  Definite Improvement (2) | 25 | 10
  Considerable Improvement (3) | 19 | 18
  Clearing (4) | 13 | 25
  Missing | 1 | 3

4. Secondary Outcome: Number of Participants With a Decrease in Signs of Psoriasis (Erythema) Scores From Baseline to Week 4
Description: Number of participants with a decrease in Signs of Psoriasis (Erythema) scores from Baseline to Week 4. Signs of Psoriasis (Erythema) are evaluated on a scale from 0 - 4 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe/Very Severe with 0 being best and 4 being worst.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat; LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Clear (0) | 5 | 4
  Almost Clear (1) | 6 | 15
  Mild (2) | 31 | 32
  Moderate (3) | 28 | 17
  Severe/Very Severe (4) | 0 | 0

5. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Scaling) Scores From Baseline to Week 4
Description: Number of participants with decrease in Signs of Psoriasis (Scaling) scores from Baseline to Week 4. Signs of Psoriasis (Scaling) are evaluated on a scale from 0 - 4 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe/Very Severe) with 0 being best and 4 being worst.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat); LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Clear (0) | 12 | 20
  Almost Clear (1) | 24 | 20
  Mild (2) | 28 | 23
  Moderate (3) | 6 | 5
  Severe (4) | 0 | 0

6. Secondary Outcome: Number of Participants With Decrease in Signs of Psoriasis (Plaque Elevation) Scores From Baseline to Week 4
Description: Number of participants with decrease in Signs of Psoriasis (Plaque Elevation) scores from Baseline to Week 4. Signs of Psoriasis (Plaque Elevation) are evaluated on a scale from 0 - 4 (0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate, 4 = Severe/Very Severe) with 0 being best and 4 being worst.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat); LOCF (Last Observation Carried Forward)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Clear (0) | 6 | 11
  Almost Clear (1) | 15 | 24
  Mild (2) | 33 | 26
  Moderate (3) | 16 | 7
  Severe/Very Severe (4) | 0 | 0

7. Secondary Outcome: Median Percent (%) Change From Baseline in % Treatable BSA (Body Surface Area) From Baseline to Week 4
Description: Median percent (%) change from baseline in % treatable BSA (Body Surface Area) from Baseline to Week 4
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat); LOCF (Last Observation Carried Forward)
Measure: Median (Standard Deviation); unit: Percent change
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
Percent change | -33.3 (31.85) | -50.0 (30.15)

8. Secondary Outcome: Mean Change From Baseline Scores for the Koo-Menter Psoriasis Index 12-item Quality of Life Questionnaire (PQOL-12) From Baseline to Week 4
Description: Mean change from baseline scores for the Koo-Menter Psoriasis Index 12-item Quality of Life Questionnaire (PQOL-12) from Baseline to Week 4. The Koo-Menter Psoriasis Index is a questionnaire with 12 questions that can be used to assess the effect that psoriasis has on a patient's overall quality of life. The questions are answered on a scale from 0 to 10 with 0 being best and 10 being worst.
Time Frame: Baseline to Week 4
Population: ITT (Intent to Treat)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
Units on a scale | -24.8 (22.81) | -27.5 (27.10)

9. Secondary Outcome: Number of Participants Who Responded to the Categories of Possible Answers to the Subject's Satisfaction Survey Question "The Treatment Program Was Easy to Follow" at Week 4
Description: Number of participants who responded to the categories of possible answers to the Subject's Satisfaction Survey question "The treatment program was easy to follow" at Week 4. Categories of possible answers include Strongly agree, Moderately agree, No opinion, Moderately disagree, and Strongly disagree.
Time Frame: Baseline and Week 4
Population: ITT (Intent to Treat)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Strongly agree | 61 | 59
  Moderately agree | 2 | 8
  No opinion | 2 | 0
  Moderately disagree | 2 | 0
  Strongly disagree | 0 | 0
  Missing | 3 | 1

10. Secondary Outcome: Number of Participants Who Responded to the Categories of Possible Answers to the Subject's Satisfaction Survey Question "I am Satisfied With my Appearance" at Week 4
Description: Number of participants who responded to the categories of possible answers to the Subject's Satisfaction Survey question "I am Satisfied with my Appearance" at Week 4. Categories of possible answers include Strongly agree, Moderately agree, No opinion, Moderately disagree, and Strongly disagree.
Time Frame: Week 4
Population: ITT (Intent to Treat)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Strongly agree | 10 | 25
  Moderately agree | 39 | 32
  No opinion | 6 | 4
  Moderately disagree | 9 | 5
  Strongly disagree | 3 | 1
  Missing | 3 | 1

11. Secondary Outcome: Number of Participants Who Responded to the Categories of Possible Answers to the Subject's Satisfaction Survey Question "I am Satisfied With the Results of This Treatment Program" at Week 4
Description: Number of participants who responded to the categories of possible answers to the Subject's Satisfaction Survey question "I am satisfied with the results of this treatment program" at Week 4. Categories of possible answers include Strongly agree, Moderately agree, No opinion, Moderately disagree, and Strongly disagree.
Time Frame: Week 4
Population: ITT (Intent to Treat)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Strongly agree | 23 | 42
  Moderately agree | 35 | 20
  No opinion | 5 | 1
  Moderately disagree | 3 | 4
  Strongly disagree | 1 | 0
  Missing | 3 | 1

12. Secondary Outcome: Number of Participants Who Responded to the Categories of Possible Answers to the Subject's Satisfaction Survey Question "I Would Use This Treatment Program Again if Recommended by the Dermatologist" at Week 4
Description: Number of participants who responded to the categories of possible answers to the Subject's Satisfaction Survey question "I would use this treatment program again if recommended by the dermatologist" at Week 4. Categories of possible answers include Strongly agree, Moderately agree, No opinion, Moderately disagree, and Strongly disagree.
Time Frame: Week 4
Population: ITT (Intent to Treat)
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants
  Strongly agree | 37 | 50
  Moderately agree | 21 | 16
  No opinion | 3 | 0
  Moderately disagree | 2 | 1
  Strongly disagree | 4 | 0
  Missing | 3 | 1

13. Secondary Outcome: Number of Participants With Tolerability Assessments Resulting in Adverse Events From Baseline to Week 4
Description: Number of participants with Tolerability Assessments resulting in Adverse Events from baseline to week 4. Tolerability assessments (Pruritus, telangiectasias, and stinging/burning) are evaluated on a scale from 0 - 3 (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) with 0 being best and 3 being worst. Skin atrophy and folliculitis are evaluated as absent or present. Changes in tolerability assessments that require a dose modification or concomitant medications/therapy are recorded as adverse events.
Time Frame: Baseline to Week 4
Population: Safety
Measure: Number; unit: participants
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Number analyzed (Participants) | 70 | 68
participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.
Arm/Group | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) | Clobex® Spray (Morning) and Vectical® Ointment (Evening)
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/68
Other Adverse Events (participants affected / at risk) | 4/70 | 0/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vectical® Ointment (Weekdays) and Clobex® Spray (Weekends) (N=70) | Clobex® Spray (Morning) and Vectical® Ointment (Evening) (N=68)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) — Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.